CLINICAL TRIAL: NCT04894162
Title: Participating in Palliative Care Research
Acronym: PiPCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: NHCT0230
Record Dates: First submitted 2021-02-18; First posted 2021-05-20 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-04

CONDITIONS: Palliative Care; Terminal Illness; Hospice Care
Keywords: research preferences
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Research questionnaire for all patients sequentially admitted to a specialist palliative care inpatient unit - 2 NHS inpatient units and 1 independent hospice.
  This is not part of standard care and data does not contribute to usual care. As such this is 'interventional' research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential recruitment of all inpatients (Other): Consecutive, eligible inpatients in a participating specialist palliative care unit will be invited to participate in the research: those who wish to participate will complete a questionnaire about research preferences.
  This is not part of standard care and results do not contribute to usual care - thus is an 'interventional' study.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Consecutive, eligible inpatients in a participating specialist palliative care unit will be invited to participate in the research: those who wish to participate will complete a research questionnaire about research preferences.

SUMMARY:
This research seeks the views of patients who are admitted to hospices and specialist palliative care units (SPCUs) regarding whether they would consider being involved in different types of clinical research. This is a questionnaire based study of inpatients in the North East of England.

The results will be used to inform healthcare professionals about the research which patients may or may not be interested in, as well as enabling future research design to be supportive of patient preferences.

Many of the interventions used within specialist palliative care lack a strong evidence base with guidelines often based on a mixture of expert opinion, anecdotal evidence or extrapolated from research in other patient groups rather than robust clinical research. Previous studies have highlighted multiple potential barriers to expanding research within the palliative care setting. Barriers include a lack of funding compared to other medical specialties and a lack of institutional capacity.

An ongoing barrier to research in this field is that the nature of the population makes patient recruitment to research challenging. This may be associated with professionals in palliative care being reluctant to ask patients if they would want to be involved in research as they feel that it would be inappropriate to potentially burden patients who are very unwell with research which is unlikely to change the disease outcome for the individual. However, many recognise that it is important to understand what patients themselves think about the potential to take part in clinical research.

Our main research question will help us to ascertain whether patients admitted under Palliative Medicine in our region would welcome the opportunity to be involved in clinical research. Previous studies have been at a single site with small numbers of patients, whereas our research will aim to recruit a larger number of patients and will be a multi-centre study involving a range of inpatient settings including an independent hospice, two National Health Service (NHS) Palliative Care Units. These centres are across the north-east region (Northumbria and Newcastle) and accept admissions from a mixture of affluent and less affluent areas. It will also involve patients with both malignant and non-malignant disease. Previous studies have not surveyed patients that were described as "too unwell", therefore as a secondary outcome we will be recording how well patients are functionally (by recording performance status- AKPS) to examine if those patients who are most unwell would still want to be involved in research. There is a gap in current knowledge of whether those patients with advanced disease and close to end of life would still find it rewarding to have the opportunity to be involved in research of some sort and whether it is fair to exclude them from being offered opportunities to be involved based on their advanced disease status.

DETAILED DESCRIPTION:
Research Question: Do patients who are cared for in specialist inpatient units in the North East of England want to take part in in research? If not, why not?

* Is there a difference in desire to participate in research between patients with malignant and non malignant disease?
* Is there a difference in desire to participate in research for patients with lower functional status?
* Is there a difference in desire to participate in research for those closer or further away from death?

From the start date of the study all consecutive admissions to the hospice or specialist palliative care units will be offered the opportunity to take part in the research study within 72 hours of their admission if they have capacity and they are under the care of the specialist palliative care team.

The opportunity to take part will be offered by a designated member of the of the multi-professional team with training in capacity assessment. This will occur at three designated times during the week to ensure both minimal disruption to patient care provision and that patients are given the opportunity to participate within 72 hours of their admission. Whilst the researchers appreciate only recruiting three times a week may miss patients with a very short length of stay it is felt that the risk of this is outweighed by reducing disruption to patient care and facilitating participation across multiple sites.

Patients will be provided with information using a patient information leaflet. This leaflet will make it clear that the decision to take part will have no impact on their usual care, and they are able to withdraw at any point in the future. The leaflet can either be read by the patient or read to the patient depending on the presence of any difficulties with reading (incl. literacy level, visual impairment and fatigue).

If the patient wishes to participate, they will be asked to sign a consent form and then given the research questionnaire to complete.

The questionnaire will be placed in a sealed envelope will be given back to a member of the healthcare team, or deposited in a collection box situated at a (manned) front desk or reception area.

Once completed consent forms and research questionnaires are received, the data will be transferred by the research team on each site to an on-site database. At this point, demographic details will be added on to the database to include age, gender, postcode, performance status and main diagnosis. The patient's NHS number will be included on the database, in order to be able to assess the patient outcome following completion of the questionnaire after 3 and 6 months. This enables the important question regarding whether the desire to participate in research changes with a shorter prognosis.

Completed research questionnaires will be gathered three times a week and stored in a locked drawer of a locked office on each research site. No patient identifiable information will be transferred between sites.

Consecutive research questionnaires for all eligible patients will be gathered. A minimum sample size of 100 patients will be recruited so that we would have a minimum ratio of events to predictor variables (age and sex) of 10, allowing us to perform meaningful analysis and minimise the risk of overfitting and type II error inflation.

Demographic data regarding the patient's underlying condition and functional status will be collected contemporaneously.

Outcome data regarding the patient's location of care will be collected at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient on a specialist palliative care unit
* Admitted in the study period.
* Over 18 years of age
* Willing to participate
* Able to complete the questionnaire (with or without support) during their admission

Exclusion Criteria:

* Lack of capacity to consent to involvement in the study
* Clinical team consider the offer of participation may cause distress or burden
* Patients not under the care of the specialist palliative care team e.g. medical borders (this exclusion criteria is only relevant to the specialist palliative care units attached to hospitals and not the hospice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients admitted consecutively to specialist palliative care inpatient units in the North east of England who wish to participate in research - binary Yes/No outcome. | 6 months
  Questionnaire study of consecutively admitted inpatients in specialist palliative care inpatient units.

SECONDARY OUTCOMES:
Proportion of patients who express a desire to participate in research who have malignant (vs non-malignant) disease. | 6 months
  Details of diagnosis (malignant or non-malignant) will be gathered to determine whether there is a difference between those with cancer and those with non-malignant disease, in relation to their preferences for research participation.
Proportion of patients who express a desire to participate in research who have an Australia-modified Karnofsky Performance Scale (AKPS) of ≥70%, between 40% and 60% and ≤30% respectively. | 6 months
  Data regarding functional status (using the Australia-modified Karnofsky Performance Scale) will be gathered to determine whether there is a difference between those with higher or lower functional scores, in relation to their preferences for research participation.
Proportion of patients who express a desire to participate in research who survive ≤1 week, ≤ 2weeks, ≤3 weeks, ≤4weeks, between 4-6 weeks, between 6-8 weeks, between 8-12 weeks, between 3-6 months and >6 months from completion of questionnaire. | 18 months from first patient recruitment
  Outcome data (regarding living at home, in care home, in hospital or death) will be gathered after 3 and 6 months following completion of the questionnaire, to determine whether there is a difference between those who have a shorter or longer prognosis, and their desire to participate in research.

CONTACTS AND LOCATIONS:
Overall Officials: Peta Heslop, Study Director — Northumbria Healthcare NHS FT - Head of R&D
Locations (3):
- United Kingdom (3):
  - Wansbeck General Hospital, Ashington
  - St Oswald's Hospice, Newcastle
  - North Tyneside General Hospital, North Shields

IPD SHARING:
Plan to Share IPD: No
Identifiable data will be kept on-site and not shared between organisations.

REFERENCES:
- [Background] Higginson IJ. Research challenges in palliative and end of life care. BMJ Support Palliat Care. 2016 Mar;6(1):2-4. doi: 10.1136/bmjspcare-2015-001091. No abstract available. PMID 26893386
- [Background] Lunder U, Sauter S, Furst CJ. Evidence-based palliative care: beliefs and evidence for changing practice. Palliat Med. 2004 May;18(4):265-6. doi: 10.1191/0269216304pm900ed. No abstract available. PMID 15198115
- [Background] Chen EK, Riffin C, Reid MC, Adelman R, Warmington M, Mehta SS, Pillemer K. Why is high-quality research on palliative care so hard to do? Barriers to improved research from a survey of palliative care researchers. J Palliat Med. 2014 Jul;17(7):782-7. doi: 10.1089/jpm.2013.0589. Epub 2014 Jun 2. PMID 24885960
- [Background] Terry W, Olson LG, Ravenscroft P, Wilss L, Boulton-Lewis G. Hospice patients' views on research in palliative care. Intern Med J. 2006 Jul;36(7):406-13. doi: 10.1111/j.1445-5994.2006.01078.x. PMID 16780445
- [Background] White C, Hardy J. What do palliative care patients and their relatives think about research in palliative care?-a systematic review. Support Care Cancer. 2010 Aug;18(8):905-11. doi: 10.1007/s00520-009-0724-1. Epub 2009 Aug 25. PMID 19705165
- [Background] Ross C, Cornbleet M. Attitudes of patients and staff to research in a specialist palliative care unit. Palliat Med. 2003 Sep;17(6):491-7. doi: 10.1191/0269216303pm785oa. PMID 14526881
- [Background] Henderson M, Addington-Hall JM, Hotopf M. The willingness of palliative care patients to participate in research. J Pain Symptom Manage. 2005 Feb;29(2):116-8. doi: 10.1016/j.jpainsymman.2004.12.001. No abstract available. PMID 15733802
- [Background] White CD, Hardy JR, Gilshenan KS, Charles MA, Pinkerton CR. Randomised controlled trials of palliative care - a survey of the views of advanced cancer patients and their relatives. Eur J Cancer. 2008 Sep;44(13):1820-8. doi: 10.1016/j.ejca.2008.05.003. Epub 2008 Jun 10. PMID 18550360
- [Background] Downing A, Morris EJ, Corrigan N, Sebag-Montefiore D, Finan PJ, Thomas JD, Chapman M, Hamilton R, Campbell H, Cameron D, Kaplan R, Parmar M, Stephens R, Seymour M, Gregory W, Selby P. High hospital research participation and improved colorectal cancer survival outcomes: a population-based study. Gut. 2017 Jan;66(1):89-96. doi: 10.1136/gutjnl-2015-311308. Epub 2016 Oct 19. PMID 27797935